CLINICAL TRIAL: NCT02261103
Title: A Multiple Dose Study With Increasing Pramipexole Doses (0.375 mg to 4.5 mg q.d.) of Oral Extended Release (ER) Tablets With a Three-way Cross Comparison of 4.5 mg Pramipexole ER q.d. Fasted Versus 4.5 mg Pramipexole ER q.d. Fed Versus 1.5 mg Pramipexole Immediate Release Tablets t.i.d. Fasted in Healthy Male Volunteers
Brief Title: Bioavailability of Increasing Pramipexole Doses of Oral Extended Release (ER) Tablets in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 248.530
Record Dates: First submitted 2014-10-09; First posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (3):
- Pramipexole IR, fasted (Active Comparator): Pramipexole immediate release (IR) tablets
  Interventions: Drug: Pramipexole IR tablets; Drug: Placebo matching Pramipexole ER tablets
- Pramipexole ER, fasted (Experimental): Pramipexole extended release (ER) tablets
  Interventions: Drug: Pramipexole ER tablets; Drug: Placebo matching Pramipexole IR tablets
- Pramipexole ER, fed (Experimental): Pramipexole extended release tablets with a high-fat meal 30 min before drug administration
  Interventions: Drug: Pramipexole ER tablets; Other: Standard high-fat breakfast

INTERVENTIONS:
Drug: Pramipexole ER tablets
  Arms: Pramipexole ER, fasted; Pramipexole ER, fed
Drug: Pramipexole IR tablets
  Arms: Pramipexole IR, fasted
Drug: Placebo matching Pramipexole ER tablets
  Arms: Pramipexole IR, fasted
Drug: Placebo matching Pramipexole IR tablets
  Arms: Pramipexole ER, fasted
Other: Standard high-fat breakfast
  Arms: Pramipexole ER, fed

SUMMARY:
The objectives of the studies are:

* To demonstrate similar total exposure between pramipexole ER fasted and pramipexole ER fed after multiple administration of the highest daily dose of 4.5 mg q.d. and to reveal any food effect leading to uncontrolled release
* To investigate the relative bioavailability of the ER-formulation of pramipexole in comparison to the IR-formulation at the highest daily dose of 4.5 mg after multiple dosing
* To demonstrate dose proportionality between the dose strengths of the pramipexole ER formulation of 0.375, 0.75, 1.5, 3.0, and 4.5 mg after multiple daily (q.d.) dosing

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study should be healthy males
* Age range from 21 to 50 years
* Body mass index (BMI) be within 18.5 to 29.9 kg/m2
* In accordance with Good Clinical Practice and the local legislation all volunteers will have given their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24:00 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (≤ one month prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on in-house trial days
* Alcohol abuse (> 40 g/day)
* Drug abuse
* Blood donation (≥ 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the clinically accepted reference range
* Excessive physical activities within the last week before the trial or during the trial
* Hypersensitivity to pramipexole, or other dopamine agonists
* Supine blood pressure at screening of systolic < 110 mmHg and diastolic < 60 mmHg

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2006-04; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ=0-24h (AUC0-24,ss) for ER | up to 23 hours after drug application on day 5
AUC0-24,ss for IR | up to 23 hours after drug application on day 5
Maximum measured concentration of the analyte in plasma at steady state (Cmax) | up to 23 hours after drug application on day 5
Area under the concentration-time curve of the analyte in plasma over the time interval 0 to 4h at steady state (AUC0-4,ss) for ER | up to 4 hours after drug application

SECONDARY OUTCOMES:
Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | up to 23 hours after drug application on day 5
Peak-Trough Fluctuation (PTF) | up to 23 hours after drug application on day 5
Time from last dosing to the maximum concentration of the analyte in plasma at steady state over a uniform dosing interval τ (tmax,ss) | up to 23 hours after drug application on day 5
Area under the concentration-time curve of the analyte in plasma over the time interval 0 to 8 h at steady state (AUC0-8,ss) | up to 8 hours after drug application
Predose concentration of the analyte in plasma at steady state immediately before administration of the next dose (Cpre,ss) | predose on days 1 to 5
Average concentration of the analyte in plasma at steady state (Cavg) | up to 23 hours after drug application on day 5
Terminal half-life of the analyte in plasma at steady state (t1/2,ss) | up to 23 hours after drug application on day 5
Mean residence time of the analyte in the body at steady state after p.o. administration (MRTpo,ss) | up to 23 hours after drug application on day 5
Apparent clearance of the analyte in plasma at steady state after extravascular multiple dose administration (CL/F,ss) | up to 23 hours after drug application on day 5
Renal clearance of the analyte at steady state determined over the dosing interval τ (CLR,ss) | up to 23 hours after drug application on day 5
Apparent volume of distribution during the terminal phase λz at steady state following extravascular administration (Vz/F,ss) | up to 23 hours after drug application on day 5
Amount of analyte that is eliminated in urine at steady state from the time point 0 to time point 24 (Ae0-24,ss) | up to 23 hours after drug application on day 5
Amount of analyte that is eliminated in urine at steady state from the time point 0 to time point 8 (Ae0-8,ss) for IR | up to 8 hours after drug application on day 5
Number of subjects with adverse events | up to 7 days after last drug administration
Number of subjects with clinically relevant changes in vital signs | up to 7 days after last drug administration
Number of subjects with clinically relevant changes in laboratory parameters | up to 7 days after last drug administration
Assessment of global tolerability by investigator on a 4-point scale | day 5 of each visit